CLINICAL TRIAL: NCT04816097
Title: Role of Prophylactic Dexamethasone Administration Before Elective Cesarean Section at Term in Reducing the Incidence of Neonatal Respiratory Distress Syndrome (A Randomized Controlled Trial)
Brief Title: Dexamethasone Before Elective Cesarean Section at Term in Reducing Neonatal Respiratory Distress Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Abass, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Steroids for lung maturity
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: C08.381.840.500.475; C08.381.840.500.737
MeSH Terms: interventions — dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Steroid Group (Active Comparator): Participants will receive 4 doses of dexamethasone 6mg IM 48h before elective CS.
  Interventions: Drug: Dexamethasone phosphate
- No Steroid Group (No Intervention): Participants will receive No treatment before elective CS.

INTERVENTIONS:
Drug: Dexamethasone phosphate — 4 doses of dexamethasone 6mg IM 48h before elective CS.
  Arms: Steroid Group

SUMMARY:
Prophylactic antenatal administration of corticosteroid enhance fetal lung maturity and reduce the probability of respiratory morbidity in preterm births.

assessment of administration of four doses intramuscular dexamethasone 48h before elective cesarean section at term in reducing the incidence of neonatal respiratory distress syndrome and NICU admission as a result

DETAILED DESCRIPTION:
Term neonates born between (37-39 wks) by elective cesarean section are likely to develop respiratory distress syndrome more than neonates born by vaginal delivery, and this risk increases for the subgroup of neonates born after elective caeserean section , i.e. before onset of labour , , with potentially severe implications The risk is decreasing with advanced gestational age and neonates born in 37 weeks are at 1.7 times more than those born at 38 weeks , which in turn are at 2.4 times more than those born at 39 weeks If the pregnant female is given four intramuscular injections of 6 mg of dexamethasone , 48 hrs before elective caesarean section decreases the neonatal respiratory morbidity. Five studies lasting between 3 to 20 years with more than 1500 patients have shown no adverse effect of single course of antenatal corticosteroid , neither through infection of the fetus or mother nor in long term neurological or cognitive effect According to Cochrane Database of Systematic Reviews 2018 , prophylactic administration of antenatal corticosteroids appeared to reduce the rate of RDS by approximately 52%. It also reduced the need for NICU admission, both due to respiratory morbidity (by approximately 58%) and for any indication. The reduction of NICU admissions due to respiratory reasons is consistent with the reduction of respiratory morbidity after corticosteroid administration

ELIGIBILITY:
Inclusion Criteria:

* Gestational age (37-39wks).
* Singleton pregnancy.
* Didn't receive any steroid treatment during pregnancy.

Exclusion Criteria:

* Undetermined gestational age
* Maternal chronic diseases (e.g: hypertension, DM-2) to avoid any side effects of steroid use and to keep the pregnant 's case from getting worse.
* Congenital fetal malformations
* Emergency CS
* Pregnant refusing to participate in the study or unable to consent

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 950 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
incidence of neonatal respiratory distress syndrome (RDS) | 1st 6 hours after delivery

SECONDARY OUTCOMES:
APGAR score | 1 min after delivery
  A: Activity/muscle tone
  0 points: limp or floppy
  1. point: limbs flexed
  2. points: active movement P: Pulse/heart rate
  0 points: absent
  1. point: less than 100 beats per minute
  2. points: greater than 100 beats per minute G: Grimace (response to stimulation, such as suctioning the baby's nose)
  0 points: absent
  1. point: facial movement/grimace with stimulation
  2. points: cough or sneeze, cry and withdrawal of foot with stimulation A: Appearance (color)
  0 points: blue, bluish-gray, or pale all over
  1. point: body pink but extremities blue
  2. points: pink all over R: Respiration/breathing
  0 points: absent
  1. point: irregular, weak crying
  2. points: good, strong cry
APGAR score | 5 min after delivery
  A: Activity/muscle tone
  0 points: limp or floppy
  1. point: limbs flexed
  2. points: active movement P: Pulse/heart rate
  0 points: absent
  1. point: less than 100 beats per minute
  2. points: greater than 100 beats per minute G: Grimace (response to stimulation, such as suctioning the baby's nose)
  0 points: absent
  1. point: facial movement/grimace with stimulation
  2. points: cough or sneeze, cry and withdrawal of foot with stimulation A: Appearance (color)
  0 points: blue, bluish-gray, or pale all over
  1. point: body pink but extremities blue
  2. points: pink all over R: Respiration/breathing
  0 points: absent
  1. point: irregular, weak crying
  2. points: good, strong cry
Rate of Neonatal intraventricular hemorrhage (IVH) | within 1st 48 hours after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Awad, Professor, Study Chair — AinSU

IPD SHARING:
Plan to Share IPD: No